CLINICAL TRIAL: NCT04288544
Title: Pilot Study "Health Promoting Effects of the Microalgae Phaeodactylum Tricornutum"
Brief Title: "Health Promoting Effects of the Microalgae Phaeodactylum Tricornutum"
Acronym: UniHoh-Algen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hohenheim (Other)
Responsible Party: Principal Investigator, Stephan C. Bischoff, MD, Professor, Professor, University of Hohenheim
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UHohenheim
Record Dates: First submitted 2020-02-21; First posted 2020-02-28 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Human Nutrition, Omega-3 Fatty Acids, Microalgae; Micronutrients
Keywords: eicosapentaenoic acid, Nutrition, micronutrients, anti-inflammatory foods, omega-3 fatty acids, microalgae
MeSH Terms: interventions — Docosahexaenoic Acids

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental: Intervention group (Active Comparator): The patients get 1x 5,3g per day the microalgae Phaeodactylum tricornutumover for two weeks.
  Interventions: Dietary Supplement: Omega-3-fatty acid capsule; Dietary Supplement: sea fish
- Omega-3 capsules (Active Comparator): The patients get one capsule per day of the Omega-3-fatty acid capsules for 2 weeks.
  Interventions: Dietary Supplement: Microalgae; Dietary Supplement: sea fish
- sea fish (facultative) (Experimental): as positive control, one portion of fish is eaten per week for 2 weeks after the Intervention of 8 weeks and 2 wash out (omega 3 must not be eaten).
  Interventions: Dietary Supplement: Microalgae; Dietary Supplement: Omega-3-fatty acid capsule

INTERVENTIONS:
Dietary Supplement: Microalgae — Open, monocentric intervention study in crossover design
  Arms: Omega-3 capsules; sea fish (facultative)
Dietary Supplement: Omega-3-fatty acid capsule — Open, monocentric intervention study in crossover design
  Arms: Experimental: Intervention group; sea fish (facultative)
Dietary Supplement: sea fish — Open, monocentric intervention study in crossover design
  Arms: Experimental: Intervention group; Omega-3 capsules

SUMMARY:
The aim of the research project is to investigate the uptake of omega-3 fatty acids into the blood plasma through the consumption of the microalgae Phaeodactylum tricornutum (PT) in a human study. In an open, crossover study, the volunteers will receive a drink enriched with the microalgae P. tricornutum or an omega-3 fatty acid preparation or (optionally) pollock for 14 days each. Since the microalgae P. tricornutum is rich in omega-3 fatty acids, the target parameter chosen is the uptake of omega-3 fatty acids in the blood plasma

DETAILED DESCRIPTION:
A large number of diet-related diseases, such as obesity, are characterized by subclinical inflammation of the body. For this reason, anti-inflammatory foods such as omega-3 fatty acids, which are found in fish and nuts, are used. However, the disadvantage of fish as a resource is its limited availability. Therefore, it is of great interest to provide a resource-saving diet that still supplies us with all macro and micro nutrients. For this reason, microalgae have become the focus of science in recent years. Microalgae not only serve as a source of protein, but also contain a large number of nutrients that could have possible physiological and preventive effects in human nutrition. These include substances from the group of carotenoids and the various polyunsaturated FS found in microalgae.

The microalgae PT is rich in omega-3 FS eicosapentaenoic acid (EPA), which is otherwise found mainly in fatty fish, and could therefore be an alternative or vegetarian source of polyunsaturated fatty acids.

Previous work by U. Neumann has shown that the microalgae P. tricornutum could be used for human nutrition. No toxic effects could be observed in vivo and the bioavailability of fatty acids and proteins could also be successfully demonstrated. In vitro experiments also showed a more anti-inflammatory, anti-oxidative and anti-proliferative effect on human blood cells. For this reason, a health-promoting effect is also possible in human nutrition, but this must be proven in human studies.

ELIGIBILITY:
Inclusion Criteria:

* Signed declaration of consent
* Willingness to follow the prescribed diet for the duration of the study
* No participation in another clinical trial (current or within the last 30 days)

Exclusion Criteria:

* Taking intestinal therapeutics, antibiotics, immunosuppressive drugs or similar (if necessary, individual case decision)
* Pregnancy/nursing period
* Relevant violations of the food protocol
* Occurrence of relevant diseases (if necessary, individual case decision)
* Revocation of consent
* Accommodation in a clinic or similar institution due to official or court order

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-25 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-09-15 (Actual)

PRIMARY OUTCOMES:
change of concentration of omega-3 fatty acids in blood plasma | Study examinations are before intervention, after 2,3,4,6,7,8, 10,11 and 12 weeks.
  concentration of fatty acids from plasma by direct transesterification and subsequent measurement on gas chromatography.

SECONDARY OUTCOMES:
change of concentration of amino acids and carotenoids (fucoxanthin) | Study examinations are before intervention, after 2,3,4,6,7,8, 10,11 and 12 weeks.
  determination of amino acids from plasma by a gas chromatography determination of carotenoids from plasma by HPLC

OTHER OUTCOMES:
change of Inflammation markers in the blood (c-reactive protein (crp) | Study examinations are before intervention, after 2,3,4,6,7,8, 10,11 and 12 weeks.
  determination of inflammation markers in serum
change of short-chain fatty acids in stool parameters | Stool samples are collected before intervention after 4,8 and 12 weeks.
  stool samples are analysed by gas chromatography (short-chain fatty acids)
change of microbiome (stool samples) | Stool samples are collected before intervention after 4,8 and 12 weeks.
  quantitative Analyse with Next-Generation Sequencing.
change of Inflammation markers in the blood like IL-6, IL-1β | study examinations are before intervention, after 2,3,4,6,7,8, 10,11 and 12 weeks.
  determination of inflammation markers in plasma with ELISA

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - lena Stiefvatter, Stuttgart
  - University of Hohenheim, Stuttgart

IPD SHARING:
Plan to Share IPD: Undecided